CLINICAL TRIAL: NCT05976763
Title: A Randomized Phase 3 Trial of Continuous vs. Intermittent Maintenance Therapy With Zanubrutinib as Upfront Treatment in Older Patients With Mantle Cell Lymphoma
Brief Title: Testing Continuous Versus Intermittent Treatment With the Study Drug Zanubrutinib for Older Patients With Previously Untreated Mantle Cell Lymphoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A052101; NCI-2023-03577 (Other: NCI Clinical Trial Reporting Program)
Record Dates: First submitted 2023-07-26; First posted 2023-08-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — zanubrutinib; Rituximab; Watchful Waiting; Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy; Endoscopy, Digestive System; Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Induction therapy (Zanubrutinib, rituximab) (Experimental): Patients receive zanubrutinib PO and rituximab IV on study. Patients undergo bone marrow biopsy and FDG PET/CT or CT throughout the trial. Patients may also undergo EDG and/or colonoscopy on study as clinically indicated. Patients may optionally undergo blood sample collection throughout the trial.
  Interventions: Drug: Zanubrutinib; Biological: Rituximab; Other: Patient Observation; Procedure: Bone Marrow Biopsy; Other: Fludeoxyglucose F-18; Procedure: Positron Emission Tomography; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Esophagogastroduodenoscopy; Procedure: Colonoscopy; Procedure: Biospecimen Collection; Other: Questionnaire Administration
- Arm A (Zanubrutinib) (Experimental): Patients receive zanubrutinib PO until first disease progression on study. Patients undergo CT or MRI or FDG PET/CT throughout the trial. Patients may optionally undergo blood sample collection throughout the trial.
  Interventions: Drug: Zanubrutinib; Other: Patient Observation; Procedure: Bone Marrow Biopsy; Other: Fludeoxyglucose F-18; Procedure: Positron Emission Tomography; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Esophagogastroduodenoscopy; Procedure: Colonoscopy; Procedure: Biospecimen Collection; Other: Questionnaire Administration
- ARM B (Observation) (Active Comparator): Patients undergo observation until first disease progression and then receive zanubrutinib PO until second disease progression on study. Patients undergo CT or MRI or FDG PET/CT throughout the trial. Patients may optionally undergo blood sample collection throughout the trial.
  Interventions: Drug: Zanubrutinib; Other: Patient Observation; Procedure: Bone Marrow Biopsy; Other: Fludeoxyglucose F-18; Procedure: Positron Emission Tomography; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Esophagogastroduodenoscopy; Procedure: Colonoscopy; Procedure: Biospecimen Collection; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Zanubrutinib — Given PO
Biological: Rituximab — Given IV
  Arms: Induction therapy (Zanubrutinib, rituximab)
Other: Patient Observation — Undergo observation
Procedure: Bone Marrow Biopsy — undergo bone marrow biopsy
Other: Fludeoxyglucose F-18 — Given IV
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: PET
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT Scan; CT Scan
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: MRI
Procedure: Esophagogastroduodenoscopy — Undergo EGD
  Other Names: EGD
Procedure: Colonoscopy — Undergo colonoscopy
Procedure: Biospecimen Collection — Undergo blood sample collection
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase III trial tests whether continuous or intermittent zanubrutinib after achieving a complete remission (CR) with rituximab works in older adult patients with mantle cell lymphoma (MCL) who have not received treatment in the past (previously untreated). Rituximab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. Zanubrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. When zanubrutinib is used in MCL, the current standard of care is to continue administering the drug indefinitely until disease progression. This continuous treatment comes with clinical as well as financial toxicity, which could be especially detrimental in older patients. For patients who achieve a CR after initial zanubrutinib plus rituximab therapy, it may be safe and equally effective to stop treatment and restart zanubrutinib upon disease progression rather than continuing indefinitely in previously untreated older adult patients with MCL.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare time to first progression or death (progression free survival [PFS]1) with continuous treatment (Arm A) and time to second progression or death (PFS2) with intermittent treatment that is restarted at first progression (Arm B).

KEY SECONDARY OBJECTIVE:

I. To compare overall survival between patients who achieve a complete remission (CR) with induction therapy subsequently treated with continuous treatment versus (vs.) intermittent treatment as part of maintenance therapy.

SECONDARY OBJECTIVES:

I. To determine overall response rate (ORR) and CR rate to induction therapy with zanubrutinib and rituximab in previously untreated MCL.

II. To determine adverse events during induction and post-induction in each study arm (Arm A and B) by Common Terminology Criteria for Adverse Events (CTCAE) 5.0.

III. To determine PFS1, event free survival (EFS) and overall survival (OS) in each study arm (A and B).

IV. To determine the overall response rate (ORR) and complete response rate (CR) after restarting zanubrutinib, following the first progression, in the intermittent treatment arm (Arm B).

V. To compare burden of symptomatic adverse events (AEs) as assessed by Patient-Reported Outcome Common Terminology Criteria for Adverse Events (PRO-CTCAE) between patients randomized to Arm A versus Arm B.

QUALITY OF LIFE PRIMARY OBJECTIVE:

I. To compare health-related quality of life (QOL) at 12 cycles post-randomization as assessed by the Functional Assessment of Cancer Therapy (FACT) Lymphoma Symptom Index-18 (FLYMSI-18) total score between patients randomized to Arm A versus Arm B.

QUALITY OF LIFE SECONDARY OBJECTIVES:

I. To compare health-related QOL at other time points as assessed by the FLYMSI-18 total score between patients randomized to Arm A versus Arm B.

II. To compare burden of symptomatic AEs as assessed by PRO-CTCAE between patients randomized to continuous (Arm A) versus intermittent (Arm B) zanubrutinib treatment.

QUALITY OF LIFE EXPLORATORY OBJECTIVES:

I. To compare the geriatric functional and cognitive PRO as assessed by Elderly Functional Index (EFLI) and Neurology (Neuro) QOL in Arm A versus Arm B.

II. To compare cognitive function at various time points as assessed by the Neuro-QOL between patients randomized to continuous (Arm A) versus intermittent (Arm B) zanubrutinib treatment.

EXPLORATORY OBJECTIVES:

I. To evaluate the completion rate of a lymphoma-specific patient assessment of life survey (PALS) with patient directed questions on life, health, and social determinants of health (SDH) and assess the impact of the survey collected data on outcomes for all enrolled patients (study arms A and B).

II. To evaluate minimal residual disease (MRD) in those patients who achieve a CR after induction therapy (arms A and B) and how detectable MRD status changes after continued therapy vs. discontinuation of therapy (i.e. arms A vs. B).

OUTLINE:

INDUCTION THERAPY: Patients receive zanubrutinib orally (PO) and rituximab intravenously (IV) on study. Patients undergo bone marrow biopsy and fluciclovine F18 (FDG) positron emission tomography (PET)/ computed tomography (CT) or CT throughout the trial. Patients may also undergo esophagogastroduodenoscopy (EGD) and/or colonoscopy on study as clinically indicated. Patients may optionally undergo blood sample collection throughout the trial.

MAINTENANCE THERAPY: Patients achieving a CR after induction therapy are randomized to 1 of 2 arms.

ARM A: Patients receive zanubrutinib PO until first disease progression on study. Patients undergo CT or magnetic resonance imaging (MRI) or FDG PET/CT throughout the trial. Patients may optionally undergo blood sample collection throughout the trial.

ARM B: Patients undergo observation until first disease progression and then receive zanubrutinib PO until second disease progression on study. Patients undergo CT or MRI or FDG PET/CT throughout the trial. Patients may optionally undergo blood sample collection throughout the trial.

After completion of study treatment, patients are followed within 30 days and every 6 months for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* • Histologically confirmed mantle cell lymphoma with cyclin D1 (BCL1) expression by immunohistochemical stains and/or t(11;14) by cytogenetics or fluorescence in situ hybridization (FISH) as confirmed by the enrolling center

  * Any stage allowed (stage I-IV)

    * Presence of measurable disease, defined as >= 1 nodal lesion that is > 1.5 cm in longest diameter or >= 1 extranodal lesion that is > 1 cm in longest diameter
    * Steroids for management of mantle cell lymphoma are allowed up to a dose of prednisone 100mg/day (or equivalent) for up to 7 days
    * No prior systemic treatment for mantle cell lymphoma
    * No prior radiation treatment for stage I MCL
    * No prior exposure to a BTK inhibitor or anti-CD20 monoclonal antibody
    * No prior stem cell transplant
    * Age >= 70 years OR age >= 60 to < 70 years with comorbidities precluding autologous stem cell transplantation (autoSCT) including at least one of the following: a) cardiac ejection fraction (EF) < 45%, b) diffusing capacity for carbon monoxide < 60% predicted; c) creatinine clearance < 70 but > 30ml/minute (min); d) Eastern Cooperative Oncology Group (ECOG) performance status of 2, which poses an unacceptable risk of toxicity for high-dose therapy and stem cell transplantation; or e) Cumulative Illness Rating Scales (CIRS) total score > 6
    * ECOG Performance Status 0-2
    * Absolute neutrophil count (ANC) >= 750/mm^3 (without growth factor support within 7 days)
    * Platelet count >= 75,000/mm^3 (or >= 50,000/mm^3 for patients with bone marrow involvement of lymphoma) without growth factor support or transfusion within 7 days
    * Creatinine clearance >= 30 mL/ min determined by either: a) Estimation using the Cockcroft-Gault equation or b) Measurement by nuclear medicine scan or 24 hour urine collection
    * Total bilirubin =< 1.5 x upper limit of normal (ULN) (unless documented Gilbert's syndrome)
    * Aspartate transferase (AST) / alanine transaminase (ALT) =< 3 x ULN
    * Patients should not be considered candidates for stem cell transplant or must have declined a stem cell transplant strategy
    * No clinically significant cardiovascular disease including the following
  * Unstable angina within 3 months before registration
  * New York Heart Association class III or IV congestive heart failure
  * History of clinically significant arrhythmias (eg, sustained ventricular tachycardia, ventricular fibrillation, torsades de pointes)
  * QT correction formula (QTcF) > 480 msecs based on Fredericia's formula
  * History of Mobitz II second-degree or third-degree heart block without a permanent pacemaker in place

    * Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
    * No active Hepatitis B or Hepatitis C infection. Patients with prior hepatitis B virus (HBV) exposure (positive HBV core antibody and/or surface antigen) are eligible if they have no detectable viral load, and are taking appropriate prophylactic antiviral therapy to prevent reactivation. Patients with history of hepatitis C virus (HCV) are eligible if they have an undetectable HCV viral load
    * Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
    * No history of severe bleeding disorder such as hemophilia A, hemophilia B, von Willebrand disease, or history of spontaneous bleeding requiring blood transfusion or other medical intervention
    * No history of stroke or intracranial hemorrhage within 6 months prior to registration
    * No disease significantly affecting gastrointestinal function such as malabsorption syndrome, resection of the stomach or small bowel, bariatric surgery procedures, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction. Patient must be able to swallow pills
    * Potential trial participants should have recovered from major surgery
    * No vaccination with a live vaccine within 35 days prior to registration
    * No hypersensitivity to zanubrutinib or rituximab or any of the other ingredients of the study drugs
    * Chronic concomitant treatment with strong inhibitors of CYP3A4 is not allowed on this study. Patients on strong CYP3A4 inhibitors must discontinue the drug for 14 days prior to registration on the study.
    * Chronic concomitant treatment with strong CYP3A4 inducers is not allowed. Patients must discontinue the drug 14 days prior to the start of study treatment
    * Avoid use of moderate CYP3A4 inhibitors, PGP inhibitors, and moderate CYP3A4 inducers
    * Archival tissue must be available for submission in all patients for histopathology review, though participation in correlative substudies is optional

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2038-08-31 (Estimated); Study Completion 2038-08-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) 1 (Arm A) | Time from randomization until the earlier of first progression or death from any cause, assessed up to 10 years
  Hazard ratios on the treatment effect will be estimated using a stratified cox proportional hazards model, stratified on age and mantle cell lymphoma (MCL) International Prognostic Index (IPI) score. The primary analysis for non-inferiority will be based on an intent-to-treat (ITT) analysis and will include all randomized patients in the analyses, regardless of eligibility or treatment status. Sensitivity analyses will also be done in an ancillary manner to evaluate and compare our endpoints using a modified ITT approach, and exclude from the analysis those classified as ineligible as well as those who withdraw right after randomization prior to any treatment/observation monitoring.
Progression-free survival (PFS) 2 (Arm B) | Time from randomization until the earlier of second progression or death from any cause, assessed up to 10 years
  Hazard ratios on the treatment effect will be estimated using a stratified cox proportional hazards model, stratified on age and MCL IPI score. The primary analysis for non-inferiority will be based on an ITT analysis and will include all randomized patients in the analyses, regardless of eligibility or treatment status. Sensitivity analyses will also be done in an ancillary manner to evaluate and compare our endpoints using a modified ITT approach, and exclude from the analysis those classified as ineligible as well as those who withdraw right after randomization prior to any treatment/observation monitoring.

SECONDARY OUTCOMES:
Overall survival (OS) (Arms A and B) | Time from randomization until death from any cause, assessed up to 10 years
  Kaplan-Meier methodology will be used to estimate the distributions of OS by treatment arm and log-rank test statistics will be used to compare these distributions between the two treatment arms. Cox Proportional Hazards models may be used to further evaluate covariates of interest with OS, including assessment of treatment effects when adjusting for other known risk factors in the model.
Incidence of adverse events | Up to 10 years
  Will be evaluated and captured using the CTCAE 5.0, where the type and severity grade of each adverse event will be collected and tabulated within each of the treatment arms. Perceived attribution to study treatment will also be captured.
  The analysis population for this secondary endpoint will include all patients who are registered and randomized on the study and receive at least one dose of study treatment. Adverse events will be monitored continuously throughout the course of the study as well as analyzed at the time of the final primary endpoint analysis.
  Summary statistics and frequency tables will be used to describe the distributions of adverse events. Rates of adverse events occurring in compared across the treatment arms with chi-squared tests Tolerability will also be evaluated, summarizing rates of dose delays or modifications, reasons patients end treatment, and time to end of active treatment.
Overall response rate (ORR, complete + partial remission) | up to 10 years
  Will be assessed using Lugano criteria. ORR to induction is defined as the number of patients with complete or partial remission at the end of induction divided by the number of patients who receive at least one dose of the induction regimen. ORR to restart of zanubrutinib is only defined for Arm B, as the number of patients with complete or partial remission after restart of zanubrutinib divided by the number of patients that restart zanubrutinib after first disease progression following randomization. The frequencies and rates of tumor response categories will be summarized by treatment arm for response to induction as well as response to restart of zanubrutinib (Arm B only). ORR to induction and ORR to restart of zanubrutinib (Arm B only) with 95% exact binomial confidence intervals will be calculated by treatment arm. To compare the association of treatment arm and ORR to induction, chi-squared or Fisher's Exact test will be used, whichever is more appropriate at final analysis.
Complete response rate (CR) | Up to 10 years
  Will be assessed using Lugano criteria. CR to induction is defined as the number of patients with complete remission at the end of induction divided by the number of eligible patients who receive at least one dose of the induction regimen. CR to restart of zanubrutinib is only defined for Arm B, as the number of patients with complete remission after restart of zanubrutinib divided by the number of eligible patients that restart zanubrutinib after first disease progression following randomization. CR to induction and CR to restart of zanubrutinib (Arm B patients only) with 95% exact binomial confidence intervals will be calculated by treatment arm. To compare the association of treatment arm and CR to induction, chi-squared or Fisher's Exact test will be used, whichever is more appropriate at the time of the final analysis.
Event-free survival (EFS) 1 | Time from randomization (Arms A and B) until the earlier of first progression, start of an alternative MCL therapy, or death from any cause, assessed up to 10 years.
  For EFS1, patients without an event will be censored at the last known clinical assessment. Any patient who goes to transplant will be censored at the last known clinical assessment prior to transplant. Kaplan-Meier methodology will be used to estimate the distribution of EFS. Cox Proportional Hazards models may be used to further evaluate covariates of interest with EFS.
Event-free survival (EFS) 2 | Time from randomization (Arm B) until the earlier of second progression, start of an alternative MCL therapy, or death from any cause, assessed up to 10 years.
  For EFS2, patients without an event will be censored at the last known clinical assessment. Any patient who goes to transplant will be censored at the last known clinical assessment prior to transplant. Kaplan-Meier methodology will be used to estimate the distribution of EFS. Cox Proportional Hazards models may be used to further evaluate covariates of interest with EFS.

CONTACTS AND LOCATIONS:
Locations (230):
- United States (230):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Tower Cancer Research Foundation, Beverly Hills, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - City of Hope at Irvine Lennar, Irvine, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital Care Center at Long Ridge, Stamford, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Emory Johns Creek Hospital, Johns Creek, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - University of Illinois, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Northwest Cancer Center - Main Campus, Crown Point, Indiana
  - Northwest Oncology LLC, Dyer, Indiana
  - Northwest Cancer Center - Hobart, Hobart, Indiana
  - Saint Mary Medical Center, Hobart, Indiana
  - Saint Catherine Hospital, Indianapolis, Indiana
  - The Community Hospital, Munster, Indiana
  - Women's Diagnostic Center - Munster, Munster, Indiana
  - Northwest Cancer Center - Valparaiso, Valparaiso, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - UI Healthcare Mission Cancer and Blood - Fort Dodge, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - HaysMed, Hays, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Freeman Physician Group of Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Alliance for Clinical Trials in Oncology, Boston, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - McLaren Cancer Institute-Central Michigan, Mount Pleasant, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - Briarcliff, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology Oncology Associates of CNY at Camillus, Camillus, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Rhode Island Hospital, Providence, Rhode Island
  - Smilow Cancer Hospital Care Center - Westerly, Westerly, Rhode Island
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - ThedaCare Regional Medical Center - Appleton, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Froedtert and MCW Moorland Reserve Health Center, New Berlin, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided